CLINICAL TRIAL: NCT06871852
Title: The Effect of a Video- and Brochure-Based Physiotherapy and Exercise Program on Migraine Symptoms, Neck Disability, Cognitive Functions, and Quality of Life in Patients with Migraine: a Randomized Controlled Trial
Brief Title: The Effect of a Video-Based Exercise Program on Migraine Symptoms
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Gulhan Yilmaz Gokmen, Assoc. Prof., Bandırma Onyedi Eylül University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-292
Record Dates: First submitted 2025-02-11; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Migraine; Exercise
Keywords: migraine; exercise; video-based; telerehabilitation
MeSH Terms: conditions — Migraine Disorders; Motor Activity

STUDY DESIGN:
Intervention Model Description: randomized controlled study (3 group)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Video-Based Intervention Group (Experimental): Group 1 - video-based physiotherapy and exercise program: Video-Based Intervention Group: Participants in this group will receive videos detailing migraine triggers, precautionary measures, and a physiotherapy and exercise program. Each exercise will be thoroughly explained by a physiotherapist in the videos, enabling participants to perform the exercises correctly by following the verbal and visual instructions. To ensure proper technique, additional video recordings will be provided to address participants' questions upon request.
  Interventions: Other: a video-based physiotherapy and exercise program.
- Brochure-Based Intervention Group (Experimental): Brochure-Based Intervention Group: Participants in this group will be provided with brochures that include information on migraine triggers, precautionary measures, and rehabilitation exercises accompanied by visual aids. The exercises will be detailed with written instructions and illustrations.
  Interventions: Other: brochure-based physiotherapy and exercise program.
- control group (No Intervention): No exercise/training will be given to the control group.

INTERVENTIONS:
Other: a video-based physiotherapy and exercise program. — Video-Based Intervention Group: Participants in this group will receive videos detailing migraine triggers, precautionary measures, and a physiotherapy and exercise program. Each exercise will be thoroughly explained by a physiotherapist in the videos, enabling participants to perform the exercises correctly by following the verbal and visual instructions.
  Arms: Video-Based Intervention Group
Other: brochure-based physiotherapy and exercise program. — Brochure-Based Intervention Group: Participants in this group will be provided with brochures that include information on migraine triggers, precautionary measures, and rehabilitation exercises accompanied by visual aids. The exercises will be detailed with written instructions and illustrations.
  Exercise Program: The exercise program will include self-massage techniques for specific muscle groups, self C1-C2 joint mobilization, cervical region exercises, cognitive exercises, and progressive relaxation exercises for the back and face.
  Arms: Brochure-Based Intervention Group

SUMMARY:
The aim of this study is to investigate the effects of a video- and brochure-based physiotherapy and exercise program on migraine symptoms, neck disability, cognitive functions, and quality of life in patients with migraine.

Hypotheses H1: The video-based physiotherapy and exercise program has an effect on migraine symptoms in patients with migraine.

H2: The video-based physiotherapy and exercise program has an effect on neck disability in patients with migraine.

H3: The video-based physiotherapy and exercise program has an effect on cognitive functions in patients with migraine.

H4: The video-based physiotherapy and exercise program has an effect on quality of life in patients with migraine.

H5: The brochure-based physiotherapy and exercise program has an effect on migraine symptoms in patients with migraine.

H6: The brochure-based physiotherapy and exercise program has an effect on neck disability in patients with migraine.

H7: The brochure-based physiotherapy and exercise program has an effect on cognitive functions in patients with migraine.

H8: The brochure-based physiotherapy and exercise program has an effect on quality of life in patients with migraine.

Participants diagnosed with migraine who meet the inclusion criteria and voluntarily agree to participate in the study will be randomly assigned to three groups using block randomization. The study will be conducted online.

Before the intervention, participants will be asked to complete the Demographic Information Form, Migraine Disability Assessment (MIDAS) Questionnaire, Mig-Scog Questionnaire, Neck Disability Index (NDI), and SF-12 Quality of Life Questionnaire via an online Google Form.

Group 1 will receive a video-based physiotherapy and exercise program. Group 2 will receive a brochure-based physiotherapy and exercise program. Group 3 will serve as the control group. Participants in the intervention groups will be instructed to perform the exercises three times per week for 12 weeks, with one session per day, consisting of 10 repetitions for each exercise.

At the end of the 12th week, all assessments will be repeated to evaluate the effects of the intervention.

DETAILED DESCRIPTION:
Migraine is commonly treated with medication; however, some patients are unable to tolerate acute and/or prophylactic medications due to side effects or contraindications associated with comorbid conditions such as myocardial disorders or asthma. The prevalence of neck pain is high among individuals with migraine, and various dysfunctions in the cervical region have been observed, including increased sensitivity of the cranio-cervical muscles, reduced force production in cervical extensor muscles, impaired performance of deep flexor muscles, decreased cervical range of motion (ROM), and hypomobility of the upper cervical segments (C1-C2).

There is increasing evidence supporting the role of physiotherapy in migraine treatment, with two primary approaches currently proposed for patient management: addressing musculoskeletal dysfunctions in the cranio-cervical region and managing postural control impairments. Furthermore, nearly 80% of migraine patients report experiencing some degree of neck pain during the migraine cycle. The prevalence of neck pain exceeds that of nausea, which is considered a diagnostic criterion for migraine. The presence of neck pain is associated with a more severe clinical presentation of migraine and may even reduce responsiveness to pharmacological treatment, thereby increasing the overall burden of the condition. Additionally, the perception of muscle tension in the neck is linked to more intense migraine attacks.

To facilitate patient adherence to exercise programs, videos and brochures are commonly used. Videos are easy to understand and can effectively simulate live demonstrations, while brochures can be tailored and customized to meet individual patient needs. Video- and brochure-based programs offer an alternative for patients who face challenges in attending in-person treatment sessions, such as those with conflicting work schedules or other barriers to participation. A review of the literature reveals a lack of studies investigating the efficacy of video- and brochure-based physiotherapy and exercise programs for migraine management.

Existing studies have primarily focused on either a single type of exercise intervention or physiotherapy techniques applied exclusively by a physiotherapist. This study aims to include exercises that migraine patients can perform independently, along with physiotherapy techniques and guidance on essential considerations, triggering factors, and recommendations for migraine management. Since migraine patients often prefer to remain indoors during episodes, accessing video-based instruction or brochures in a comfortable environment may facilitate treatment adherence.

The objective of this study is to examine the effects of a video- and brochure-based self-administered physiotherapy and exercise program on migraine symptoms, neck disability, cognitive functions, and quality of life in individuals with migraine.

ELIGIBILITY:
Inclusion Criteria:

1. Migraine has been diagnosed by a specialist physician
2. Between the ages of 18 and 65
3. Volunteering to participate in the study
4. To be able to answer surveys sent from a smart phone or computer

Exclusion Criteria:

1. Having secondary diseases such as morbid obesity, blood pressure, diabetes
2. Any other neurological or psychiatric disorder
3. Severe cervical disc herniation or radiculopathy
4. Receiving any other treatment for migraine during the study (except medication)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
The Migraine Disability Assessment (MIDAS) | baseline - after 3 months
  The Migraine Disability Assessment (MIDAS) questionnaire is a brief, self-administered tool designed to measure headache-related disability over a three-month period. It consists of five items that assess the number of days, in the past 3 months, of activity limitations due to migraine. Higher scores indicate greater disability. The MIDAS questionnaire has been shown to be internally consistent, highly reliable, valid, and correlates with physicians' clinical judgment. Consequently, it is widely used in clinical research as a standard assessment tool.
The Migraine-Specific Cognitive Assessment (Mig-SCog) | baseline - after 3 months
  The Migraine-Specific Cognitive Assessment (Mig-SCog) is a self-administered questionnaire developed in 2011 by Gil-Gouveia and colleagues to assess and monitor cognitive symptoms during migraine attacks. The scale consists of nine Likert-type items, each scored from 0 to 2, with a total score ranging from 0 to 18; higher scores indicate a greater frequency of cognitive symptoms. The first three items assess attention, processing speed, and orientation; items four and five evaluate planning and attention; items six and seven pertain to language; and items eight and nine focus on naming. Thus, the Mig-SCog primarily examines executive functions (attention, planning, and orientation) and language (naming and verbal fluency), which are the areas most commonly reported as problematic by patients during migraine attacks. A high Mig-SCog score indicates a high frequency of cognitive symptoms.

SECONDARY OUTCOMES:
The Neck Disability Index (NDI) | Baseline- after 3 months
  The Neck Disability Index (NDI) is a self-report questionnaire designed to assess how neck pain affects a patient's daily life. Developed in 1989 by Howard Vernon, it is widely used in both clinical and research settings. The NDI consists of 10 items, each scored on a scale from 0 to 5, with higher scores indicating greater disability. The total score can range from 0 to 50 and is often expressed as a percentage. Interpretation of the scores is as follows:
  0-4: No disability 5-14: Mild disability 15-24: Moderate disability 25-34: Severe disability 35-50: Complete disability The NDI has been shown to have good reliability and validity in various studies. A change of 5 points is considered the minimal clinically important difference, indicating a meaningful change in a patient's condition. The questionnaire typically takes between 3 to 7.8 minutes to complete.
The Short Form-12 (SF-12) | baseline - after 3 months
  The Short Form-12 (SF-12) is a concise health survey derived from the SF-36, designed to assess overall health status efficiently. Developed in 1995, the SF-12 has been validated in various languages, including Turkish. Studies have found that the SF-12's psychometric properties are comparable to those of the SF-36. The Physical Component Score (PCS) is derived from subdomains such as general health, physical functioning, role-physical, and bodily pain, while the Mental Component Score (MCS) is obtained from subdomains including social functioning, role-emotional, mental health, and vitality.
The Exercise Adherence Rating Scale (EARS) | baseline - after 3 months
  The Exercise Adherence Rating Scale (EARS) is a valid and reliable tool developed by Newman and colleagues to assess exercise adherence behavior. It provides a simple, standardized, and reliable evaluation of adherence to prescribed home exercises, facilitating the development and assessment of interventions that promote long-term self-management for both the prevention and treatment of chronic conditions. The EARS consists of three sections:
  Section A: Comprising six items that can be adapted to personal needs; this section is not included in the scale scoring.
  Section B: The core part of the scale, which cannot be adapted to personal needs, describes how the recommended home exercises are performed.
  Section C: Evaluates the reasons for adherence or non-adherence to the recommended home exercises.
  The items of the measurement tool are scored between 1 and 4. Scores of 1 and 2 indicate irrelevance, 3 and 4 indicate interest. A high EARS score indicates good compliance with exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- Bandirma Onyedi Eylul University, Bandırma, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No